CLINICAL TRIAL: NCT03164837
Title: Safety and Diagnostic Performance of 68Gallium-labeled NOTA-RM26 PET/CT in Prostate Cancer Patients
Brief Title: 68Ga-NOTA-RM26 PET/CT in Prostate Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM021; ZIAEB000073 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 68Ga-NOTA-RM26

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-RM26 PET/CT (Experimental): The patients were injected with 111-148 MBq of 68Ga-NOTA-RM26 in one dose intravenously and underwent PET/CT scan 15-30 min later.
  Interventions: Drug: 68Ga-NOTA-RM26

INTERVENTIONS:
Drug: 68Ga-NOTA-RM26 — Single-dose 68Ga-NOTA-RM26 were injected into the patients before the PET/CT scans.

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-RM26 in prostate cancer patients. A single dose of 111-148 Mega-Becquerel (MBq) 68Ga-NOTA-RM26 will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
The gastrin-releasing peptide receptor (GRPR), also known as bombesin receptor subtype II (BB2), is a member of the G protein-coupled receptor family of bombesin receptors. GRPR is over-expressed in various types of human tumors including prostate cancer. RM26, a GRPR antagonist with high affinity, was discovered by peptide backbone modification of bombesin analogues.To target gastrin-releasing peptide receptor in neoplastic cells of human prostate cancer, peptide NOTA-RM26 was synthesized with a PEG3 linker between NOTA and RM26, and then labeled with 68Ga. An open-label whole-body PET/ CT study was designed to investigate the safety and dosimetry of 68Ga-NOTA-RM26 and to assess its clinical diagnostic value in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of primary prostate cancer having a prostate neoplasm identified by ultrasound or MRI, being diagnosed by needle biopsy as having prostate cancer, having undergone whole-body bone scanning, and being able to provide basic information and sign the written informed consent form.

Exclusion Criteria:

* The exclusion criteria included claustrophobia, kidney or liver failure, and inability to fulfill the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-RM26 in prostate cancer | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in prostate cancer will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, M.D.,PhD., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China